CLINICAL TRIAL: NCT04062617
Title: Complications of Endoscopic Retrograde Cholangio-Pancreatography (ERCP) - an Indian Perspective
Brief Title: Cmplications of ERCP
Acronym: C-ERCP
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: AMRI Hospital, Salt Lake, Kolkata, India (Unknown)
Responsible Party: Principal Investigator, Kshaunish Das, Professor, Division of Gastroenterology, School of Digestive and Liver Disease, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC/2018/567
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Complication of ERCP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a form of endoscopy where a Side-viewing endoscope is introduced into the duodenum, following which instruments are passed into bile or pancreatic ducts, to allow their radiological visualisation by injecting contrast medium and/or perform various therapeutic procedures, e.g., removal of bile duct stone. It is a complex endoscopic procedure with long learning curve and has number of complications which can even be life-threatening. Since its introduction in 1968, ERCP has become a widely used endoscopic procedure for a variety of disorders. Endoscopic biliary sphincterotomy was first reported in 1974. ERCP at its inception was predominantly a diagnostic procedure, however over the past decade its predominantly carried out for therapeutic indications because of the availability of other imaging techniques, such as abdominal Ultrasound (US), Computed Tomography (CT), Magnetic resonance cholangiopancreatography (MRCP), Endoscopic Ultrasound (EUS) that provide detailed diagnostic information and thus allowing appropriate selection of patients for therapeutic ERCP. Complications are expected to occur in a proportion of patients undergoing ERCP, even when performed by endoscopists with significant expertise in the procedure. A number of patient-related and technique-related factors are known to increase the risk of complication. ERCP requires sedation and therefore has in addition a risk of anaesthesia related adverse events. Most of the complications post-ERCP are apparent during the first 6 hours after the procedure. There are no large scale study evaluating the complications of ERCP in Indian or even Asian population. In an attempt to address this deficit we will be conducting a dual centre prospective study to look at the incidence of various ERCP-related complications. Proposed study will be done in both a tertiary care public academic centre and a tertiarycare private hospital. Both have specialised and well equipped department to carry out ERCP procedures and evaluate and manage complications if any.

DETAILED DESCRIPTION:
INTRODUCTION:

Endoscopic retrograde cholangiopancreatography (ERCP) is a form of endoscopy where a Side-viewing endoscope is introduced into the duodenum, following which instruments are passed into bile or pancreatic ducts, to allow their radiological visualisation by injecting contrast medium and/or perform various therapeutic procedures, e.g., removal of bile duct stone. It is a complex endoscopic procedure with long learning curve and has number of complications which can even be life-threatening.(1) . Since its introduction in 1968, ERCP has become a widely used endoscopic procedure for a variety of disorders (2).

Endoscopic biliary sphincterotomy was first reported in 1974(3). ERCP at its inception was predominantly a diagnostic procedure, however over the past decade its predominantly carried out for therapeutic indications (4-5) because of the availability of other imaging techniques, such as abdominal Ultrasound (US), Computed Tomography (CT), Magnetic resonance cholangiopancreatography (MRCP), Endoscopic Ultrasound (EUS) that provide detailed diagnostic information and thus allowing appropriate selection of patients for therapeutic ERCP. Complications are expected to occur in a proportion of patients undergoing ERCP, even when performed by endoscopists with significant expertise in the procedure. A number of patient-related and technique-related factors are known to increase the risk of complication (6). ERCP requires sedation and therefore has in addition a risk of anaesthesia related adverse events (7). Most of the complications post-ERCP are apparent during the first 6 hours after the procedure (8). Thus patients require careful monitoring during this phase to detect symptoms or signs suggesting adverse events. Table 1 below sums up the complications related to ERCP that has been reported in various studies. (9,10,11,12,13- 21) . Table 1: Complications of ERCP Related to pancreaticobiliary instrumentation Pancreatitis Bleeding Infection

Related to technical issue with endoscopy Electrosurgical hazards:

Thermal injury: perforation Inadequate cautery: Bleeding Air insufflation: Post ERCP pain Contrast allergy Perforation

Related to anesthesia Cardiopulmonary complication:

Aspiration Hypoxemia Cardiac dysrhythmia Rare complications Gallstone ileus Colonic perforation Liver abscess splenic/hepatic/vascular trauma Pneumothorax Gas embolism Impaction of retrieval basket Biloma Multiple studies have evaluated the incidence of post ERCP complications (9,10,11,12) .

Prospective surveys from single referral centres ensure the highest accuracy but are unlikely to be representative of the frequency and severity of unfavourable events in day-to-day practice. By comparison, prospective multi-centre studies involving centres with different volumes of activity and operators with various degrees of expertise more reliably reflect the general effectiveness and safety of ERCP in the community (10,12). There are no large scale study evaluating the complications of ERCP in Indian or even Asian population. In an attempt to address this deficit we will be conducting a dual centre prospective study to look at the incidence of various ERCP-related complications.

Proposed study will be done in both a tertiary care public academic centre and a tertiarycare private hospital. Both have specialised and well equipped department to carry out ERCP procedures and evaluate and manage complications if any.

REVIEW OF LITERATURE:

ERCP is used to diagnose and intervene therapeutically in various pancreatico-biliary disorders in a minimally invasive manner. But to acquire competence a minimum of 180 procedures is required for a trainee in diagnostic and therapeutic ERCP, defined by deep cannulation of bile duct in 70 to 80 % of cases.(22) ERCP has a wide variety of indications.

ERCP is generally indicated in as per guidelines published by American Society of Gastrointestinal Endoscopy.(23)

1. The jaundiced patient suspected of having biliary obstruction (appropriate therapeutic manoeuvres should be performed during the procedure).
2. The patient without jaundice whose clinical and biochemical or imaging data suggest pancreatic duct or biliary tract disease.
3. Evaluation of signs or symptoms suggesting pancreatic malignancy when results of direct imaging (eg, EUS, US, CT, magnetic resonance imaging [MRI]) are equivocal or normal.
4. Evaluation of pancreatitis of unknown etiology.
5. Preoperative evaluation of the patient with chronic pancreatitis and/or pseudocyst.
6. Evaluation of the sphincter of Oddi by manometry. Empirical biliary sphincterotomy without sphincter of Oddi manometry is not recommended in patients with suspected type III sphincter of Oddi dysfunction.
7. Endoscopic sphincterotomy:

   7.1. Choledocholithiasis. 7.2. Papillary stenosis or sphincter of Oddi dysfunction. 7.3. To facilitate placement of biliary stents or dilation of biliary strictures.

   7.4. Sump syndrome. 7.5. Choledochocele involving the major papilla. 7.6. Ampullary carcinoma in patients who are not candidates for surgery 7.7. Facilitate access to the pancreatic duct.
8. Stent placement across benign or malignant strictures, fistulae, postoperative bile leak, or in high-risk patients with large unremovable common duct stones.
9. Dilation of ductal strictures.
10. Balloon dilation of the papilla.
11. Nasobiliary drain placement.
12. Pancreatic pseudocyst drainage in appropriate cases. M. Tissue sampling from pancreatic or bile ducts.
13. Ampullectomy of adenomatous neoplasms of the major papilla.
14. Therapy of disorders of the biliary and pancreatic ducts.
15. Facilitation of cholangioscopy and/or pancreatoscopy. It is generally recommended that patients not undergo routine pre-procedure laboratory testing, chest radiography, or electrocardiography prior to endoscopic procedures.

(24) Instead, pre procedure testing should be used selectively based on the patient's medical history, physical examination findings, and procedural risk factors. Since ERCP carries an approximate 5 percent risk of major complications, including acute pancreatitis, bleeding, sepsis, and perforation, we typically obtain laboratory tests prior to the procedure if an intervention is anticipated (such as sphincterotomy) and blood tests that have not been obtained as part of the patient's prior evaluation. Such tests include a complete blood count and prothrombin time/international normalised ratio. A consensus panel introduced a standardised, outcome-based set of definitions and grading system for the major complications of ERCP and endoscopic sphincterotomy.(9) These are noted in Table 2 and 3.

The overall specific complications (ie, pancreatitis, bleeding, sepsis, and perforation) varies from 5 to 10 percent in various studies. In a prospective study of total 2347 patients , complications occurred in 229 (9.8%) patients.(10) In a summary of 21 studies involving 16,855 patients between 1987 and 2003, specific complications totalled 1154 (6.9 percent), with 55 deaths (0.33 percent).(11) Mild-tomoderate events occurred in 872 patients (5.2 percent), and severe events in 282 (1.7 percent). Among 12,973 patients enrolled in 14 prospective studies, non specific complications totalled 173 (1.3 percent), with nine deaths (0.07 percent)(11) Despite technological progress and recommendations of scientific societies, the incidence of complications and procedure-related mortality does not appear to have decreased over time. One possible reason is that ERCP has become a primarily therapeutic procedure. In a single center Finnish study with over 1200 ERCPs performed between 2002 and 2009, the overall complication and mortality rates were 11 and 0.4 percent, respectively.

(25)

PANCREATITIS:

It is the most common complication after ERCP with most studies demonstrating rates of 1.5 to 6 percent. Table 4 demonstrates the complication rates noted in major studies assessing complication rates of ERCP done over past 20 years. Most of the cases are mild to moderate in severity. Table 5 demonstrates incidence of post ERCP pancreatitis based on their severity. The various risk factors for pancreatitis implicated in various Sphincter of Oddi dysfunction (SOOD), younger age, precut sphincterotomy, difficult cannulation, number of pancreatic contrast injection, pancreas divisum, failed clearance of biliary stone, prior post ERCP pancreatitis, female sex, normal serum bilirubin, absence of chronic pancreatitis, placement of stent and ASA score III-IV(10,26,27,28,29)

BLEEDING:

It is the second most common complication post ERCP in most studies. Bleeding was the most feared complication when therapeutic biliary endoscopy was first introduced. Because of advances in equipment and experience, it has become a relatively uncommon complication of endoscopic retrograde cholangiopancreatography (ERCP), and it is mostly observed after sphincterotomy.(22) In a review of 21 studies of over 16,000 patients undergoing ERCP, there were a total of 226 bleeding episodes (1.3 percent), with eight deaths (0.05 percent).(11) Bleeding was severe in 66 of the 226 episodes (29 percent). Table 6 enlists the major studies evaluating rate of Post ERCP bleeding. As a general rule, sphincterotomy is contraindicated in patients with severe coagulation disorders, such as patients with advanced liver disease, in patients with hematologic diseases, and in patients with disorders of hemostasis, such as hemophilia and von Willebrand disease.

SEPTIC COMPLICATIONS:

Septic complications of ERCP include ascending cholangitis, liver abscess, acute cholecystitis, infected pancreatic pseudocyst, infection following perforation of a viscus, and less commonly, endocarditis/endovasculitis(30) Ascending cholangitis: In the setting of ERCP, it is most often due to incomplete drainage of an infected and obstructed biliary system. Table 7 demonstrates incidence of cholangitis in various studies. Failure to achieve drainage of an obstructed biliary system is the most important predictor of post-ERCP biliary sepsis. Acute Cholecystitis: Acute cholecystitis following ERCP or percutaneous transhepatic biliary drainage may be more common than once appreciated, and must be distinguished from cholangitis. The incidence of acute cholecystitis in most large series having an incidence ≤0.5 percent.Table 8 lists the 2 major series evaluating the same. The pathogenesis may be related to the introduction of non-sterile contrast media into a poorly emptying gallbladder and/or mechanical or inflammatory obstruction of the cystic duct by an endoprosthesis, malignancy, or gallstone. Acute cholecystitis following ERCP should be suspected in patients who develop tenderness localised in the right upper quadrant and have thickening of the gallbladder wall and pericholecystic fluid on ultrasonography or computed tomography

PERFORATION:

Perforation is one of the most feared complications of endoscopic retrograde cholangiopancreatography. The Stapfer classification is most commonly used and is based on the mechanism, anatomical location, and severity of the injury that may predict the need for surgical intervention.(33)

* Type I: Free bowel wall perforation
* Type II: Retroperitoneal duodenal perforation secondary to periampullary injury
* Type III: Perforation of the pancreatic or bile duct
* Type IV: Retroperitoneal air alone In a case series of 44 post-ERCP perforations, 30 (68 percent) were retroperitoneal duodenal perforations, which usually occur as a result of a sphincterotomy that extends beyond the intramural portion of bile duct.(34) In a single-center series, 79 post-ERCP perforations were diagnosed: seven perforations were type I, 54 were type II, nine were type III, six were type IV, and three were hypopharyngeal or esophageal. While most patients with Type II perforations were medically managed, four patients from this group (7 percent) required surgical intervention.(13)Table 8 below demonstrates the rate of post ERCP perforation in various studies over the years. In another study, the incidence of perforation following ERCP was approximately 0.4 percent, with a mortality rate of approximately 7 to 8 percent.Type I perforations accounted for 25 percent of perforations, type II for 46 percent, type III for 22 percent, and type IV for 3 percent (35)

RARE COMPLICATIONS:

A number of less common adverse events have also been described including cardiopulmonary complications, contrast allergy, impaction of a retrieval basket, and numerous other events reported in only small numbers of patients or individual case reports.

These unusual adverse events, which may be difficult to manage, can be associated with significant morbidity and mortality. Uncommon complications of ERCP have been described in several large studies. Miscellaneous complications occurred in 25 of 2347 cases (~1 percent) in a prospective series of patients who underwent biliary sphincterotomy 5. Six of these were cardiopulmonary events, which were fatal in three patients. In a systematic review of 14 prospective studies including a total of 12,973 patients, there were a total of 173 miscellaneous complications (1.3 percent) and nine deaths (0.07 percent)(13) Anaphylactic reactions to contrast agents used during ERCP are rare.(14) Nevertheless, a history of sensitivity to iodine contrast or drug should always be considered in the preprocedure assessment and in the informed consent process. Electrocautery can influence implantable devices such as pacemakers and defibrillators.

Although most modern pacemakers are unaffected by electrocautery, cardiac arrhythmias can develop if a monopolar current passes through the pacemaker or the heart. The risk is greater for implantable cardioverter-defibrillators since electrocautery may trigger their activation. As a result, the American Society for Gastrointestinal Endoscopy Technology Assessment Committee recommends that implantable cardioverter-defibrillators be deactivated during endoscopic electrosurgery.(15) Opacification of the portal vein has been described following sphincterotomy.(16) Accidental cannulation of the hepatic artery following needle-knife sphincterotomy has also been reported.(17) Filling of portal, arterial, or lymphatic vessels has potential risks, including sepsis, air embolism, bleeding, and thrombosis. Furthermore, failed prompt recognition of contrast in vascular structures may be a source of confusion leading to prolongation of the procedure, thereby further increasing the risk of complications. As an example, an opacified portal vein may be misinterpreted as an incompletely filled bile duct. Insertion of a stent into the portal vein may further worsen the consequences. Cases of air embolism have been reported following upper and lower gastrointestinal endoscopy, although most described cases have been related to ERCP. In a review including 40 cases of systemic air embolism following an endoscopic procedure, 24 patients (60 percent) underwent ERCP (18) Hemorrhage following endoscopic sphincterotomy usually occurs in the duodenal lumen arising from the actual sphincterotomy site. In rare cases intraperitoneal hemorrhage has been described from injury to the spleen, liver, or abdominal vessels. Splenic injury is more commonly caused by colonoscopy, but it has also been reported following ERCP.(19) Previous abdominal surgery with adhesion formation is recognized as a risk factor; concomitant liver laceration has also been reported (20,21) Pneumothorax, pneumomediastinum, and pneumoperitoneum have been reported secondary to gastrointestinal perforation, including perforation following endoscopic sphincterotomy. However, pneumothorax has also been described during diagnostic upper endoscopy and during ERCP without perforation (25) Such cases are due to a rise in airway and intra alveolar pressure and the rupture of pulmonary blebs. Impaction of a Dormia basket around a large calculus was a feared complication of bile duct extraction prior to the introduction of mechanical lithotripsy. Despite the availability of lithotripsy, cases are still reported. Usually the basket becomes trapped at the ampulla within the intraduodenal portion of the common bile duct. Once the basket impaction has occurred, the first and common alternative is mechanical lithotripsy. (38) TABLE 2 - CLASSIFICATION OF COMPLICATIONS OF ERCP TABLE 3 - GRADING OF ERCP RELATED COMPLICATIONS TABLE 4 - INCIDENCE OF POST ERCP PANCREATITIS Site Focal Occuring At Point Of Endoscopic Contact Nonspecific Occuring In Organ Not Traversed/Treated Timing Immediate Occuring During Ercp Early Evident Within Recovery Period Delayed Within 30 Days Criteria for severity Length of stay/others Mild Less than 4 nights Moderate 4 to 10 nights Severe More than 10 nights, icu admission or surgery STUDY DIAGNOSTIC/ THERAPEUTIC ERCP NUMBER OF PATIENTS INCIDENCE Freeman et al 1996 (10) Endoscopic biliary sphincterotomy 2347 patients 5.4% Loperfido et al 1998 (12) Therapeutic ERCP 1827 patients 1.6% Rabenstein et al 2000 (26) Endoscopic sphincterotomy 438 patients 4.3% Freeman et al 2001(27) Diagnostic and therapeutic ERCP 1963 patients 6.7% Andriulli et al 2007 (11) (META-ANALYSIS) Diagnostic and therapeutic ERCP 16,855 patients 3.47% TABLE 5: INCIDENCE OF POST ERCP PANCREATITIS BASED ON SEVERITY TABLE 6: INCIDENCE OF POST ERCP BLEEDING TABLE 7 : INCIDENCE OF POST ERCP CHOLANGITIS +/- CHOLECYSTITIS TABLE 8 : INCIDENCE OF POST ERCP CHOLECYSTITIS MILD MODERATE SEVERE Freeman et al (10) 41.7% 51.2% 7.1%% Andriulli et al 2007 (11) (META-ANALYSIS) 44.8% 43.8% 11.4% STUDY DIAGNOSTIC/ THERAPEUTIC ERCP NUMBER OF PATIENTS INCIDENCE Freeman et al 1996 (10) Endoscopic biliary sphincterotomy 2347 patients 2.0% Loperfido et al 1998 (12) Therapeutic ERCP 1827 patients 0.76% Andriulli et al 2007 (11) (META-ANALYSIS) Diagnostic and therapeutic ERCP 16,855 patients 1.3% STUDY DIAGNOSTIC/ THERAPEUTIC ERCP NUMBER OF PATIENTS INCIDENCE Freeman et al 1996 (10) Endoscopic biliary sphincterotomy 2347 patients 1.0% Andriulli et al 2007 (11) (META-ANALYSIS) Diagnostic and therapeutic ERCP 16,855 patients 1.44% (cholecystitis and/or cholangitis) William et al 200731 Diagnostic and therapeutic ERCP 5264 patients 1.0% Kager L M et al32 Diagnostic and therapeutic ERCP 193 patients 3.4% STUDY DIAGNOSTIC/ THERAPEUTIC ERCP NUMBER OF PATIENTS INCIDENCE Freeman et al 1996(10) Endoscopic biliary sphincterotomy 2347 patients 0.5% Masci et al 2001 (29) Diagnostic and therapeutic ERCP 2103 patients 0.20% TABLE 9 : INCIDENCE OF POST ERCP PERFORATION STUDY DIAGNOSTIC/ THERAPEUTIC ERCP NUMBER OF PATIENTS INCIDEN CE Stafler et al, 2000 (33) 1993 to 1998 1417 patients 1.0 Masci et al, 2001(29) 1997 to 1998 2103 patients 0.57% Fatima et al, 2007 (36) 1994 to 2004 12,427 patients 0.61% Andriulli et al 2007 (11) (Metaanalysis) 1977-2006 16,855 patients 0.6% Motomura et al, 2014 (37) 2008 to 2013 2674 patients 0.22%

REFERENCES

1. ASGE Standards of Practice Committee, Chandrasekhara V, Khashab MA, et al. Adverse events associated with ERCP. Gastrointest Endosc 2017; 85:32.
2. McCune, WS, Shorb, PE & Moscovitz, H. Endoscopic cannulation of the ampulla of Vater: a preliminary report. Ann Surg 1968; 167: 752-6
3. Kawai, K, Akasaka, Y, Murakami, K, Tada, M, Kohill, Y & Nakajima, M. Endoscopic sphincterotomy of the ampulla of Vater. Gastrointest Endosc 1974; 20: 148-51
4. Chutkan R K et al. Endoscopic Retrograde Cholangiopancreatography (ERCP) : core curriculum. Gastrointest Endosc. 2006 Mar;63(3):361-76
5. ASGE Training committee, Jorgensen J et al. Endooscopic Retrograde Cholangiopancreatography (ERCP) : core curriculum. Gastrointest Endosc. 2016 Feb; 83(2):279-89
6. Analysis of 59 ERCP lawsuits; mainly about indications Cotton, Peter B. Gastrointestinal Endoscopy , Volume 63 , Issue 3 , 378 - 382
7. Zakeri N, Coda S et al. Risk factors for endoscopic sedation reversal events: a five-year retrospective study. Frontline Gastroenterol. 2015 Oct;6(4):270-277.
8. Ho KY, Montes H et al. Features that may predict hospital admission following outpatient therapeutic ERCP. Gastrointest Endosc. 1999 May;49(5):587-92.
9. Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991;37(3):383
10. Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996;335(13):909.
11. Andriulli A, Loperfido S, Napolitano G, et al. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol 2007; 102:1781.
12. Loperfido S, Angelini G, Benedetti G, et al. Major early complications from diagnostic and therapeutic ERCP: a prospective multicenter study. Gastrointest Endosc 1998; 48:1.
13. Kumbhari V, Sinha A, Reddy A, et al. Algorithm for the management of ERCP-related perforations. Gastrointest Endosc 2016; 83:934
14. Draganov PV, Forsmark CE. Prospective evaluation of adverse reactions to iodine containing contrast media after ERCP. Gastrointest Endosc 2008; 68:1098
15. Petersen BT, Hussain N, Marine JE, et al. Endoscopy in patients with implanted electronic devices. Gastrointest Endosc 2007; 65:561.
16. Huibregtse K, Gish R, Tytgat GN. A frightening event during endoscopic papillotomy. Gastrointest Endosc 1988; 34:67.
17. Gottschalk U, Morgenstern C, Kadow K. Accidental cannulation of the hepatic artery following needle-knife sphincterotomy. Z Gastroenterol 2007; 45:702.
18. Voigt P, Schob S, Gottschling S, et al. Systemic air embolism after endoscopy without vessel injury - A summary of reported cases. J Neurol Sci 2017; 376:93.
19. Gaffney RR, Jain V, Moyer MT. Splenic Injury and ERCP: A Possible Risk for Patients with Advanced Chronic Pancreatitis. Case Rep Gastroenterol 2012; 6:162.
20. Wu WC, Katon RM. Injury to the liver and spleen after diagnostic ERCP. Gastrointest Endosc 1993; 39:824.
21. Lo AY, Washington M, Fischer MG. Splenic trauma following endoscopic retrograde cholangiopancreatography (ERCP). Surg Endosc 1994; 8:692.
22. Jowell PS, Baillie J, Branch MS, Affronti J, Browning CL, Bute BP . Quantitative assessment of procedural competence. A prospective study of training in endoscopic retrograde cholangiopancreatography. Ann Intern Med. 1996;125(12):983.
23. ASGE Standards of Practice Committee, Early DS, Ben-Menachem T, Decker GA et al. Appropriate use of GI endoscopy.. Gastrointest Endosc. 2012 Jun;75(6):1127-31
24. ASGE Standards of Practice Committee, Pasha SF, Acosta R, Chandrasekhara V, Chathadi KV, Eloubeidi MA, Fanelli R, Faulx AL, Fonkalsrud L, Khashab MA, Lightdale JR, Muthusamy VR, Saltzman JR, Shaukat A, Wang A, Cash B. Routine laboratory testing before endoscopic procedures. Gastrointest Endosc. 2014 Jul;80(1):28-33. Epub 2014 May 15.
25. A. Siiki, A. Tamminen, T. Tomminen, P. Kuusanmäki Ercp Procedures In A Finnish Community Hospital: A Retrospective Analysis Of 1207 Cases Scandinavian Journal Of Surgery 101: 45-50, 2012
26. Rabenstein T, Schneider HT, Bulling D, Nicklas M, Katalinic A, Hahn EG, Martus P, Ell C Analysis of the risk factors associated with endoscopic sphincterotomy techniques: preliminary results of a prospective study, with emphasis on the reduced risk of acute pancreatitis with low-dose anticoagulation treatment Endoscopy. 2000;32(1):10.
27. Freeman ML, DiSario JA, Nelson DB, Fennerty MB, Lee JG, Bjorkman DJ, Overby CS, Aas J, Ryan ME, Bochna GS, Shaw MJ, Snady HW, Erickson RV, Moore JP, Roel JP Risk factors for post-ERCP pancreatitis: a prospective, multicenter study. Gastrointest Endosc. 2001;54(4):425
28. Cheng CL, Sherman S, Watkins JL, Barnett J, Freeman M, Geenen J, Ryan M, Parker H, Frakes JT, Fogel EL, Silverman WB, Dua KS, Aliperti G, Yakshe P, Uzer M, Jones W, Goff J, Lazzell-Pannell L, Rashdan A, Temkit M, Lehman GA Risk factors for post-ERCP pancreatitis: a prospective multicenter study.Am J Gastroenterol. 2006;101(1):139
29. Masci E, Toti G, Mariani A, Curioni S, Lomazzi A, Dinelli M, Minoli G, Crosta C, Comin U, Fertitta A, Prada A, Passoni GR, Testoni PA Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. Am J Gastroenterol. 2001;96(2):417
30. ASGE Standards of Practice Committee, Chandrasekhara V, Khashab MA, et al. Adverse events associated with ERCP. Gastrointest Endosc 2017; 85:32.
31. Williams EJ, Taylor S, Fairclough P, Hamlyn A, Logan RF, Martin D, Riley SA, Veitch P, Wilkinson ML, Williamson PR, Lombard M. Risk factors for complication following ERCP; results of a large-scale, prospective multicenter study. Endoscopy. 2007 Sep;39(9): 793-801.
32. Kager LM1, Sjouke B, van den Brand M, Naber TH, Ponsioen CY. The role of antibiotic prophylaxis in endoscopic retrograde cholangiopancreatography; a retrospective singlecenter evaluation.Scand J Gastroenterol. 2012
33. Stapfer M, Selby RR, Stain SC, et al. Management of duodenal perforation after endoscopic retrograde cholangiopancreatography and sphincterotomy. Ann Surg 2000; 232:191.
34. Polydorou A, Vezakis A, Fragulidis G, et al. A tailored approach to the management of perforations following endoscopic retrograde cholangiopancreatography and sphincterotomy. J Gastrointest Surg 2011; 15:2211.
35. Vezakis A, Fragulidis G, Polydorou A. Endoscopic retrograde cholangiopancreatographyrelated perforations: Diagnosis and management. World J Gastrointest Endosc 2015; 7:1135.
36. Fatima J, et al Pancreaticobiliary and duodenal perforations after periampullary endoscopic procedures: diagnosis and management. Arch Surg. 2007 May;142(5):448-54; discussion 454-5.
37. Motomura Y et al Immediate detection of endoscopic retrograde cholangiopancreatography-related periampullary perforation: fluoroscopy or endoscopy? World J Gastroenterol. 2014 Nov 14;20(42):15797-804
38. Mutignani et al. Novel Methods of Management of Trapped Dormia Baskets in the Pancreatic and Biliary Ducts. Endoscopy 1997; 29(2): 129-130D

ELIGIBILITY:
Inclusion Criteria:

* Those more than or equal to 12 years of age undergoing diagnostic or therapeutic ERCP between 1st August 2018 to 31st July 2019 either for the first time or after a previous failed cannulation attempt

Exclusion Criteria:

* Surgically altered anatomy of Upper GI tract
* Failure of endoscopist to reach second part of duodenum due to pyloroduodenal obstruction despite endoscopic attempts to relieve the obstruction (e.g., balloon dilatation of stricture).
* Those undergoing side-viewing endoscopy only with or without ampullary biopsy
* Those undergoing stent removal without any biliary/pancreatic endotherapy
* Repeat biliary endotherapy (e.g., stent exchange, second attempt at difficult stone removal) without pancreatic endotherapy
* Repeat pancreatic endotherapy without biliary endotherapy
* Immunodeficiency (primary or secondary)
* Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals referred for diagnostic or therapeutic ERCP
Sampling Method: Probability Sample
Enrollment: 929 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
To evaluate incidence of complications of diagnostic and therapeutic Endoscopic Retrograde Cholangiopancreatography (ERCP) | 30 days
  An unplanned event attributable to the ERCP procedure that requires the patient to be admitted to hospital, or to stay longer than expected, or to undergo other interventions:
  * Within 30 days of procedure
  * We do not count in complication statistics any deviation that occurs during a procedure that is not obvious to the patient afterwards, and does not require unplanned admission.

SECONDARY OUTCOMES:
To identify possible risk factors for these complications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- School of Digestive and Liver Diseases (SDLD), IPGME & R, Kolkata, Kolkata, India

IPD SHARING:
Plan to Share IPD: No